CLINICAL TRIAL: NCT03180151
Title: The Effect of Corticotomy in En-mass Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Ali Habiballah Hassan, Professor in orthodontic department, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 078-16
Record Dates: First submitted 2016-12-25; First posted 2017-06-08 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Accelerate Tooth Movement
Keywords: corticotomy; enmass retraction; mini implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthodontic tooth movement group (No Intervention): This is the control group in which pateints will be treated by conventional orthodontic treatment and extraction of premolars without piezotome
- Corticotomy assisted orthodontic group (Experimental): This is the study group in which patients will be treated by conventional orthodontic treatment aided by corticotomy procedure perfumed by using a piezotome.(piezotome assisted orthodontic tooth movement)
  Interventions: Procedure: piezotome assisted orthodontic tooth movement

INTERVENTIONS:
Procedure: piezotome assisted orthodontic tooth movement — Surgical procedure
  1. After local anesthesia, vertical interproximal incisions will be done under the interdental papilla, on the labial aspect of upper arch using a blade No. 15.
  2. The incisions will be kept minimal.
  3. The incisions go though the periosteum, which permit the blade to reach to the alveolar bone.
  4. A Piezo surgical knife will be used to make the cortical alveolar incision through the gingival incisions to a depth of approximately 3mm.
  5. As we will not use bone graft so we don't need use suturing after cortication.
  6. We give patient antibiotic and analgesic cover.
  Other Names: corticotomy assisted tooth movement
  Arms: Corticotomy assisted orthodontic group

SUMMARY:
* To compare patients who will undergo orthodontics treatment involving upper premolar extraction for space of time whether with or without corticotomy by Piezotome.
* Assess the safety of both methods of retraction in regard to the quality of the surrounding periodontium and roots of anterior teeth.
* Monitor postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* On the basis of the diagnosis of the malocclusion, individuals who have Class I and Class II malocclusions and requiring extraction of premolars and retraction of anterior teeth will be selected (maxillary/mandibular or both).
* Good oral hygiene, healthy gingiva and no evidence of bone loss as seen in radiograph.
* Healthy systemic conditions.
* No previous orthodontic treatment.
* Patient needs to be in permanent dentition (hence, we need to define their age range).

Exclusion Criteria:

* Patient with systemic disease.
* Patient having any signs of active periodontal disease.
* Patients on long-term corticosteroid therapy.
* Persons taking medications that slows down bone metabolism.
* Craniofacial anomalies.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
rate of tooth movement per time | 4 months

IPD SHARING:
Plan to Share IPD: Undecided
After publication, data can be shared with others upon request via email to the corresponding author.

REFERENCES:
- [Derived] Hatrom AA, Howait MS, Zawawi KH, Al-Turki GA, Alansari RA, Almehayawi NF, Alammari SH, Mohammed RA, Hassan AH. Pulp volume changes after piezocision-assisted tooth movement: a randomized clinical trial. BMC Oral Health. 2021 Jan 13;21(1):28. doi: 10.1186/s12903-020-01382-2. PMID 33435897